CLINICAL TRIAL: NCT07244341
Title: A Phase 1, Multicenter Trial Evaluating the Safety, Tolerability, and Efficacy of Valemetostat (DS-3201) in Combination With Darolutamide in Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: A Study of Valemetostat (DS-3201b) in Combination With Darolutamide in Metastatic Castration Resistant Prostate Cancer (mCRPC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS3201-343; 2025-522512-16-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Metastatic Castration Resistant Prostate Cancer; DS-3201; Valemetostat; Darolutamide; mCRPC
MeSH Terms: interventions — darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Dose Escalation) (Experimental): Participants will receive valemetostat at escalating doses in combination with darolutamide.
  Interventions: Drug: Valemetostat; Drug: Darolutamide
- Part 2 (Dose Expansion) (Experimental): Participants will receive valemetostat at 2 or more dose levels in combination with darolutamide.
  Interventions: Drug: Valemetostat; Drug: Darolutamide

INTERVENTIONS:
Drug: Valemetostat — Dose Escalation Part: Valemetostat will be administered at escalating doses. Dose Expansion Part: Valemetostat will be administered at 2 or more dose levels.
  Other Names: DS-3201
Drug: Darolutamide — Dose Escalation Part: Darolutamide will be administered at a standard dose. Dose Expansion Part: Darolutamide will be administered at a standard dose.
  Other Names: NUBEQA

SUMMARY:
This study will assess the safety and tolerability of valemetostat in combination with darolutamide in participants with Metastatic Castration Resistant Prostate Cancer (mCRPC).

ELIGIBILITY:
Key Inclusion Criteria:

The clinical site will screen for the full inclusion criteria per protocol.

1. Adult males ≥18 years of age at the time the ICF is signed (Please follow local regulatory requirements if the legal age of consent for trial participation is >18 years old).
2. Histologically confirmed adenocarcinoma of the prostate. Cases exhibiting neuroendocrine differentiation are eligible for enrollment, except those with a diagnosis of pure small cell carcinoma, which is excluded.
3. Evidence of disease progression as per the PCWG3 modified RECIST v1.1 criteria.
4. Evidence of metastatic disease as confirmed by radiographic imaging (CT, MRI, or bone scan).
5. Ongoing androgen deprivation at time of enrollment.

   • For participants currently being treated with luteinizing hormone-releasing hormone agonists or antagonists, therapy must have been initiated at least 4 weeks prior to enrollment and treatment must be continued throughout the trial.
6. Baseline PSA expression level of ≥2 ng/mL, according to a documented testing result.
7. Prior therapy with an Androgen Receptor Pathway Inhibitors (ARPI).
8. ECOG PS of 0 or 1 assessed no more than 28 days prior to enrollment.
9. Is willing and able to provide adequate fresh or archival tumor samples with sufficient quantity and tissue quality. A mandatory newly obtained pretreatment biopsy is required, if not clinically contraindicated and at an acceptable risk as determined by the investigator. If newly obtained tissue samples are not possible to obtain, archival tissue obtained from a lesion not previously irradiated and collected after the most recent prior therapy is acceptable.
10. A male participant capable of producing sperm is eligible to participate if he agrees to the following during the intervention period and for at least the time needed to eliminate each trial intervention. The length of time required to continue contraception after the last dose for each trial intervention is 3 months.

    * Must not freeze or donate sperm starting at screening and throughout the Treatment Period, and for at least 3 months after the final trial intervention administration.

Note: Preservation of sperm should be considered before enrollment in this trial.

• Adhere to either of the following contraception methods:

* True abstinence from penile-vaginal intercourse, when this is in line with the preferred and usual lifestyle of the participant, OR
* Uses a penile/external condom when having penile-vaginal intercourse with an NPOCBP, PLUS partner use of an additional contraceptive method, as a condom may break or leak Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical trials. If the contraception requirements in the local label for any trial interventions are more stringent than those above, the local label requirements are to be followed.

Key Exclusion Criteria:

The clinical site will screen for the full exclusion criteria per protocol.

1. Prior treatment with any epigenetic agents including but not limited to EZH1, EZH2, EZH1/2, or PRC2 inhibitors.
2. Has a super scan as seen in the baseline bone scan. A super scan is defined as an intense symmetric activity in the bones and diminished renal parenchymal activity on baseline bone scan, such that the presence of additional metastases in the future could not be evaluated.
3. Clinically active brain metastases, spinal cord compression, or leptomeningeal carcinomatosis, defined as untreated or symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms.
4. Uncontrolled or significant cardiovascular disease,
5. Prior malignancy, active within the previous 3 years except for locally curable cancers that have been apparently cured or successfully resected, such as basal or squamous cell carcinoma, superficial bladder cancer, carcinoma in situ of the stomach, or carcinoma in situ of the breast.
6. Has active or uncontrolled HBV infection.
7. Has active or uncontrolled HCV infection.
8. Has active or uncontrolled HIV infection.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The trial will enroll adult male participants (aged ≥18 years) with a confirmed diagnosis of mCRPC.
Enrollment: 60 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of participants with Dose-Limiting Toxicities (DLTs) | Day 1 up to Day 28
  A DLT is defined as any Treatment Emergent Adverse Event (TEAE) not attributable to disease or disease-related processes, environmental factors, unrelated trauma, etc, that occurs during the DLT evaluation period (Day 1 to Day 28) and is Grade ≥3.
Part 1 and 2: Number of Participants Experiencing a Treatment Emergent Adverse Event (TEAE) | From Screening up to approximately 5 years
  TEAEs are defined as those Adverse Events (AEs) with start or worsening date during the on-treatment period (from the first dose date of trial intervention to 30 days after the last dose date of trial intervention).

SECONDARY OUTCOMES:
Prostate-Specific Antigen (PSA) 50 Response Rate | From Screening up to approximately 5 years
  PSA50 response rate is defined as the percentage of participants who achieved a decline in PSA percent change from baseline by at least 50%, with a consecutive confirmation assessment at least 3 weeks later per the PCWG3 modified RECIST v1.1 criteria.
Prostate-Specific Antigen (PSA) 90 Response Rate | From Screening up to approximately 5 years
  PSA90 response rate is defined as the percentage of participants who achieved a decline in PSA percent change from baseline by at least 90%, with a consecutive confirmation assessment at least 3 weeks later per the PCWG3 modified RECIST v1.1 criteria.
Prostate-Specific Antigen (PSA) Nadir Response Rate | From Screening up to approximately 5 years
  PSA nadir response rate is defined as the proportion of participants who achieve a PSA level of ≤ 0.2 ng/mL at any time during the Treatment Period.
Radiographic Progression-Free Survival (rPFS) | From Screening up to approximately 5 years
  rPFS is defined as the time (month) from the start date of trial intervention to the earlier date of the first objective documentation of radiographic disease progression as assessed by the investigator based on the PCWG3 modified RECIST v1.1 criteria or death due to any cause.
Overall Survival (OS) | From Screening up to approximately 5 years
  OS is defined as the time (month) from the start date of trial intervention to the date of death due to any cause.
Time to PSA Progression | From Screening up to approximately 5 years
  Time to PSA progression is defined as the time interval from the start date of trial intervention to PSA progression, per the PCWG3 modified RECIST v1.1 criteria. PSA progression is defined as:
  * A ≥25% increase and an absolute increase of ≥2 ng/mL from the nadir, confirmed by a second PSA measurement obtained at least 3 weeks later, in participants who experience a decline in PSA from baseline; OR
  * A ≥25% increase and an absolute increase of ≥2 ng/mL from baseline, occurring beyond 12 weeks from treatment initiation, in participants who do not experience a PSA decline from baseline.
Objective Response Rate (ORR) | From Screening up to approximately 5 years
  ORR is defined as the proportion of participants with measurable disease who achieved a BOR of confirmed CR or confirmed PR as assessed by the investigator according to the PCWG3 modified RECIST v1.1 criteria.
Time to First SSRE (symptomatic bone fractures, spinal cord compression, surgery, or radiation to the bone, whichever is first) | From Screening up to approximately 5 years
  Time to first SSRE (symptomatic bone fractures, spinal cord compression, surgery, or radiation to the bone, whichever is first) is defined as the time interval from the start date of trial intervention to the date of the first observed SSRE.
Total and Unbound Plasma Concentration of Valemetostat in Combination with Darolutamide | Cycle 1: Day 1, Day 8, Day 15. Cycles 2-5: Day 1 (Each cycle is 28 days)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - NEXT Oncology, San Antonio, Texas
  - Virginia Cancer Specialists (NEXT Virginia), Fairfax, Virginia
- Japan (3):
  - Kobe City Med Cen Gen Hosp., Kobe
  - Cancer Institute Hospital of JFCR, Kōtoku
  - Toho University Sakura Medical Center, Sakura-shi

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/